CLINICAL TRIAL: NCT04427917
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF MULTIPLE ORAL DOSES OF PF-06835919 IN HEALTHY ADULT JAPANESE PARTICIPANTS
Brief Title: Study of Multiple Oral Doses of PF-06835919 in Healthy Adult Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C1061010; 2020-000218-13 (EudraCT Number); JAPANESE BRIDGING (Other: Alias Study Number)
Record Dates: First submitted 2020-05-12; First posted 2020-06-11 (Actual); Results first posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-03

CONDITIONS: Healthy
Keywords: NASH, KHK, PF-06835919, Japanese
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — PF-06835919

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, randomized, double-blind, sponsor-open, placebo-controlled study in healthy adult Japanese participants.
Who Masked: Participant, Investigator
Masking Description: double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PF-06835919 (Experimental)
  Interventions: Drug: PF-06835919
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06835919 — PF-06835919 300 mg repeated doses
  Arms: PF-06835919
Drug: Placebo — Placebo repeated doses
  Arms: Placebo

SUMMARY:
This is a Phase 1 study to evaluate the safety, tolerability, and pharmacokinetics of multiple oral doses of PF-06835919 in healthy adult Japanese participants.

A total of approximately 8 healthy participants will be enrolled in this study. Participants will be randomized to 2 groups to receive PF-06835919 or placebo treatment with a randomization ratio of 3:1.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants must be 18 to 55 years of age, inclusive, at the time of signing the ICD.
2. A Japanese participant is defined as having 4 biological Japanese grandparents who were born in Japan.
3. Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiovascular tests.
4. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
5. BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
6. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
3. History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, HBcAb or HCVAb. Hepatitis B vaccination (positive HBsAb) is allowed.
4. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
5. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention (Refer to Section 6.5 for additional details).
6. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
7. A positive urine drug test.
8. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest: If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
9. Baseline 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTc interval >450 msec, complete LBBB, signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate corrected using the Fridericia method (QTcF) and the resulting QTcF should be used for decision making and reporting. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
10. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * AST or ALT level ≥1.25 × ULN;
    * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.
11. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
12. Use of tobacco- or nicotine-containing products in excess of the equivalent >5 cigarettes/day or 2 chews of tobacco per day.
13. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
14. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
15. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1061010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were screened within 28 days of the first dose of study intervention. Eligible participants were admitted to the Clinical Research Unit.
Pre-assignment Details: A total of 8 healthy participants were enrolled in this study. Participants were randomized to 2 groups to receive PF-06835919 or placebo treatment with a randomization ratio of 3:1.
Groups:
- Placebo Daily (QD): Participants received matching placebo at approximately 0800 hours (plus or minus 2 hours), approximately 20 minutes prior to the start of breakfast on Days 1-7.
- PF-06835919 300 mg Daily (QD): Participants received PF-06835919 300 mg daily at approximately 0800 hours (plus or minus 2 hours), approximately 20 minutes prior to the start of breakfast on Days 1-7.
Period: Overall Study
Arm/Group | Placebo Daily (QD) | PF-06835919 300 mg Daily (QD)
Started | 2 | 6
Completed | 2 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who randomly assigned to study intervention and received at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06835919 300 mg Daily (QD) | Placebo Daily (QD) | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 2 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs , and TEAEs Leading to Participant Discontinuation From Study
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An serious adverse event (SAE) was defined as an AE: 1. resulting in death, 2. was life-threatening, 3. required inpatient hospitalization or prolongation of existing hospitalization, 4. resulted in persistent disability, 5. was a congenital anomaly/birth defect, or considered to be an important medical event. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug.
Time Frame: Baseline (Day 1) to follow-up (Day 42)
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Daily (QD) | PF-06835919 300 mg Daily (QD)
Number analyzed (Participants) | 2 | 6
Participants
  Participants with adverse events | 0 | 3
  Participants with serious adverse events | 0 | 0
  Participants discontinued from study due to adverse events | 0 | 0

2. Primary Outcome: Number of Participants With Clinical Laboratory Findings of Potential Clinical Importance
Description: To determine if there were any clinically significant laboratory abnormalities, haematological (hemoglobin, hematocrit, red blood cell count, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils and lymphocytes), clinical chemistry (blood urea nitrogen, glucose [fasting], calcium, sodium, potassium, chloride, bicarbonate, alanine aminotransferase, aspartate aminotransferase, total bilirubin, alkaline phosphatase, uric acid, albumin, total protein) and urinalysis (pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin) tests were assessed. Each parameter was evaluated against commonly used and widely accepted criteria.
Time Frame: Day 1 to Day 10
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Daily (QD) | PF-06835919 300 mg Daily (QD)
Number analyzed (Participants) | 2 | 6
Participants | 0 | 0

3. Primary Outcome: Number of Participants With ECG Data of Potential Clinical Concern
Description: ECG endpoints (QTcF, PR and QRS) meeting the criteria of potential clinical concern were summarized by treatment using categories as defined: 1.maximum post-dose QTcF ≤450msec, 450 - ≤480msec, 480 - ≤500msec and >500msec; 2. PR max. ≥300ms; 3. QRS max. ≥140ms.
Time Frame: Day 1 to Day 10
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Daily (QD) | PF-06835919 300 mg Daily (QD)
Number analyzed (Participants) | 2 | 6
Participants
  PR Interval Value ≥ 300 msec | 0 | 0
  QRS Duration Value ≥140 msec | 0 | 0
  QTcF Interval Value ≤450 msec | 2 | 6
  450 msec<QTcF Interval Value ≤480 msec | 0 | 0
  480 msec<QTcF Interval Value ≤500 msec | 0 | 0
  QTcF Interval Value >500 msec | 0 | 0

4. Primary Outcome: Number of Participants/Subjects With Vital Signs Data of Potential Clinical Concern
Description: Single supine blood pressure and pulse measurements meeting the criteria of potential clinical concern were summarized by treatment using categories as defined: 1. Systolic Blood Pressure (BP) min. <90mm Hg; 2. Diastolic BP min. <50mm Hg; 3. Supine pulse rate min. <40 bpm, max. >120 bpm.
Time Frame: From Study Day 1 up tp Study Day 10
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Daily (QD) | PF-06835919 300 mg Daily (QD)
Number analyzed (Participants) | 2 | 6
Participants
  Systolic BP < 90mm Hg | 0 | 0
  Diastolic BP < 50mm Hg | 0 | 0
  Supine Pulse Rate<40bpm or >120bpm | 0 | 0
  Standing pulse rate<40bpm or >140bpm | 0 | 0

5. Primary Outcome: Summary of Maximum Plasma Concentration (Cmax) of PF-06835919 on Day 1 and Day 7
Description: Cmax was defined as maximum observed plasma concentration.
Time Frame: Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16 on Day 1 and Day 7
Population: All participants who received at least 1 dose of PF-06835919 and who have at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | PF-06835919 300 mg Daily (QD)
Number analyzed (Participants) | 6
microgram per milliliter (mcg/mL)
  Day 1 | 23.39 (14)
  Day 7 | 30.49 (10)

6. Primary Outcome: Summary of Area Under the Plasma Concentration-Time Curve Over Dosing Interval (AUCtau) of PF-06835919 on Day 1 and Day 7
Description: AUCtau was defined as area under the plasma concentration-time curve over dosing interval.
Time Frame: Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16 on Day 1 and Day 7
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | PF-06835919 300 mg Daily (QD)
Number analyzed (Participants) | 6
mcg*hr/mL
  Day 1 | 169.3 (22)
  Day 7 | 230.9 (20)

7. Primary Outcome: Summary of Time for Maximum Observed Concentration (Tmax) of PF-06835919 on Day 1 and Day 7
Description: Tmax was defined as Time for maximum observed concentration of PF-06835919.
Time Frame: Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16 on Day 1 and Day 7
Population: All participants who received at least 1 dose of PF-06835919 and who had at least 1 of the PK parameters of interest calculated.
Measure: Median (Full Range); unit: hours
Arm/Group | PF-06835919 300 mg Daily (QD)
Number analyzed (Participants) | 6
hours
  Day 1: Tmax | 0.834 [0.500 to 2.00]
  Day 7: Tmax | 0.750 [0.500 to 1.08]

8. Primary Outcome: Summary of Terminal Half-life (t1/2) of PF-06835919 on Day 7
Description: t1/2 was defined as terminal half-life.
Time Frame: Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16 on Day 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-06835919 300 mg Daily (QD)
Number analyzed (Participants) | 6
hours | 14.62 (2.944)

ADVERSE EVENTS:
Time Frame: From Study Day 1 up to Study Day 42
Description: Same event may appear as adverse event (AE) and serious AE, what is presented as distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set included all participants who were randomized and received at least 1 confirmed dose of investigational product.
Arm/Group | Placebo Daily (QD) | PF-06835919 300 mg Daily (QD)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 0/2 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Daily (QD) (N=2) | PF-06835919 300 mg Daily (QD) (N=6)
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Weight increased (Investigations) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT04427917/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT04427917/SAP_001.pdf